CLINICAL TRIAL: NCT02020343
Title: Insulin Resistance in the Control of Intestinal Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Professor, University of Missouri-Columbia
Other Study IDs: 1208668
Record Dates: First submitted 2013-12-13; First posted 2013-12-24 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Insulin Resistance; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be collected for future determination of genotypes that impact taste senstivity
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy: Not insulin resistant
  Interventions: Behavioral: taste tests
- Insulin resistant: Insulin resistant by IVGTT
  Interventions: Behavioral: taste tests
- Type 2 diabetics: Type 2 diabetics
  Interventions: Behavioral: taste tests

INTERVENTIONS:
Behavioral: taste tests — Subjects undergo "sham feeding" in which they take a bit of food, chew it and spit it out. This test should engage sensory mechanisms which may affect intestinal signaling.

SUMMARY:
America's preferential consumption of high-fat/high-sugar foods is a driving force in the current epidemic of obesity and insulin resistance. Recent scientific observations suggest that the taste of food may play a role in how the body processes the food eaten in a meal. The intestine may play a central role in all aspects of dietary fat metabolism, from initial encounter with taste buds in the mouth to eventual triglyceride (TG) storage in the body.

The investigators hypothesize that elevated blood fats in insulin resistance are a result of elevated intestinal-TG secretion and poor communication of this organ to the rest of the body after meals.

In this study, meal feeding and sensory studies will be performed to determine whether the mechanism of taste-associated intestinal signaling leads to higher levels of blood fats after meals in 24 healthy, insulin resistant and type 2 diabetic subjects. Individuals will consume special meals the night before the tests and participate in sensory tests in the morning to analyze the effect of taste.

The goal of this work is to understand how insulin resistance may cause impaired signaling between the taste buds and the intestine to result in an elevation in blood lipids, which increases the risk for other chronic diseases. This study will generate data for a future study to understand how diabetes treatment affects this process.

DETAILED DESCRIPTION:
Subjects will participate in two screening visits to determine insulin resistance status and then participate in a single in-patient, clinical research center test.

There are no drugs used in this study. The goal is to test the physiological response to eating.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects (age 18-50y) will be categorized as:

* lean/insulin sensitive (IS) (n=8, BMI </= 24 kg/m2 and SI ≥ 2.5 min-1 10-4 * per uU/mL)
* overweight/obese IS (n=8, BMI 26-35 and SI >2.5 min-1 10-4 * per uU/mL)
* overweight/obese insulin resistant (n=8, BMI 26-35 and SI <2.5 min-1 10-4 * per uU/mL).

Overweight/obese insulin resistant subjects will have a family history of diabetes as defined as at least one parent or grandparent with type 2 diabetes, or at least one other family member with type 2 diabetes.

* Type 2 diabetic patients (BMI 26-35, and OGTT 2h glucose >/= 140 mg/dL.

Exclusion Criteria:

* BMI over 35 kg/m2: We felt it prudent to limit the additional variability that could be caused by morbid obesity (and by diabetes), given the early stages of this research area.
* Unusual eating habits (dietary fat< 30% or >40% of energy, skipping breakfast, day-long fasting, or allergies to milk). Habitual food intake can influence taste acuity and milk is used in the formulas to dissolve the isotopes.
* Uncontrolled hypertension, or occasional or regular smoker, use of supplements or medications that interfere with lipid, protein, or carbohydrate metabolism or impact taste. For example, the hypertensive drugs thiazides or the supplement chondroitin sulfate or niacin, can be associated with impaired glucose tolerance. ACE inhibitors and beta-blockers and smoking can affect taste. Use of insulin in the case of type 2 diabetics.
* Pregnancy (urine test), breastfeeding, or anemia (CBC with diff): Limitations of blood that can be drawn. Postmenopausal women frequently have increases in blood lipids since lack of estrogen influences lipid metabolism.
* Alcohol intake: Males >140 g/week, females > 70 g/week. Excess EtOH increases lipid synthesis and secretion in the liver and whether it also has an impact on intestinal TG metabolism is unknown.
* Fasting plasma TG >300 mg/dL. Extreme hypertriglyceridemia could be due to either elevations in VLDL or chylomicrons, either of which would impair our ability to resolve dietary metabolic processes.
* Exclude those who need to consume acetaminophen-containing medications on a regular basis. Acetaminophen is administered with meals to assess gastric emptying.
* Postmenopausal women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, insulin resistant and type 2 diabetic subjects.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Meal triglyceride (TG) absorption | Change in plasma TG concentrations over 24 hr after meals and in response to an acute sensory stimulus
  In vivo measurement of meal TG absorption is made using stable isotope administration into sequential meals (lunch and dinner) and analysis of plasma samples by GS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Derived] Jacome-Sosa M, Hu Q, Manrique-Acevedo CM, Phair RD, Parks EJ. Human intestinal lipid storage through sequential meals reveals faster dinner appearance is associated with hyperlipidemia. JCI Insight. 2021 Aug 9;6(15):e148378. doi: 10.1172/jci.insight.148378. PMID 34369385